CLINICAL TRIAL: NCT03463759
Title: Pro-Nociceptive and Anti-Nociceptive Mechanisms Across an Episode of Recurrent Low Back Pain
Brief Title: Pain Inhibition and Facilitation in Recurrent Low Back Pain
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Megan McPhee, PhD Fellow, Aalborg University
Other Study IDs: N-20170034
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Low Back Pain; Healthy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent Low Back Pain Patients: Participants experiencing a current episode of their recurrent non-specific low back pain at the time of recruitment.
- Healthy Volunteers: Participants matched in age and gender to one of the recurrent low back pain patients, with no significant past low back pain, chronic pain or other relevant medical disorders.

SUMMARY:
This study evaluates psychophysical measures of pain inhibition and facilitation, along with cortical responses to different sensory stimuli, in patients with recurrent low back pain and matched healthy individuals.

DETAILED DESCRIPTION:
Pain inhibitory and facilitatory mechanisms have been suggested to play a role in the development of persistent low back pain; however, there is still debate on when changes in these mechanisms occur. Similarly, evoked cortical responses can reflect neuroplastic changes in pain processing regions, which are also thought to play a role in the transition to persistent pain, but there is also debate on when these neuroplastic changes develop relative to low back pain. Therefore, this study will use patients with an intermediary clinical pain state, recurrent low back pain, and matched healthy control participants, to investigate within and between subject differences in pain inhibitory, facilitatory and neuroplastic mechanisms.

ELIGIBILITY:
Inclusion:

* Healthy men and women
* Aged 18-60 years
* No previous back pain OR >1 previous episode of low back pain in past 12 months
* No current back pain OR Pain in the region posteriorly between the inferior border of the 12th rib and the lower gluteal fold (low back pain) at time of recruitment lasting >24 hours
* Able to speak, read and understand English

Exclusion:

* Pregnancy
* First episode of low back pain
* Low back pain associated with menstruation
* Chronic low back pain (continuous pain episode for >3 months)
* Currently seeking active treatment for low back pain
* Red flags symptoms
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Current or previous neurologic, musculoskeletal, mental, or other illnesses which may affect the trial
* Current or previous chronic or recurrent pain condition other than low back pain
* Current regular use of analgesic or other medication which may affect the trial
* Lack of ability to cooperate
* Recent history of acute pain particularly in the lower limbs (unless related to LBP)
* Abnormally disrupted sleep in 24 hours preceding experiment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Population recruited from university, college, and wider Aalborg community
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Day 0 vs. Day 28
  Pressure pain threshold (kPa) as test stimulus before compared to during a pressure conditioning stimulus on the lower leg
Temporal Summation of Pain | Day 0 vs. Day 28
  Pain rating (VAS) change over a series of 10 repeated mechanical stimuli

SECONDARY OUTCOMES:
Pressure Pain Thresholds | Day 0 vs. Day 28
  Threshold of pain detection (kPa) with handheld algometry over the low back and distant sites
Thermal Pain Thresholds | Day 0 vs. Day 28
  Hot and cold pain detection thresholds (degrees)
Two Point Discrimination | Day 0 vs. Day 28
  The smallest distance (mm) for which two separate points can be distinguished over the low back
Proprioceptive Weighting | Day 0 vs. Day 28
  Center of pressure displacement during 1-minute of quiet standing
Sensory Evoked Potentials | Day 0 vs. Day 28
  EEG signals recorded in response to laser and electrical stimuli applied to the back

OTHER OUTCOMES:
Affective Regulation | Day 0 vs. Day 28
  Pressure pain ratings pre, during and post affective image set
Attentional Regulation | Day 0 vs. Day 28
  Pressure pain ratings pre, during and post computerised attention-demanding task

CONTACTS AND LOCATIONS:
Overall Officials: Megan E McPhee, BPhty MSc, Principal Investigator — Aalborg University
Locations (1):
- CNAP, SMI, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McPhee ME, Graven-Nielsen T. Positive affect and distraction enhance whereas negative affect impairs pain modulation in patients with recurrent low back pain and matched controls. Pain. 2022 May 1;163(5):887-896. doi: 10.1097/j.pain.0000000000002442. PMID 34382603